CLINICAL TRIAL: NCT03043105
Title: Thalidomide, Cyclophosphamide and Prednisone in Newly Diagnosed Multicentric Castleman's Disease: a Prospective, Single-center, Single-arm, Phase-II Pilot Trial
Brief Title: TCP Regimen in Newly Diagnosed MCD:a Prospective, Single-center, Single-arm, Phase-II Pilot Trial
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Jian Li, Associated professor in hematology, Peking Union Medical College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZS-1159
Record Dates: First submitted 2017-01-31; First posted 2017-02-03 (Estimated); Results first posted 2020-04-16 (Actual); Last update posted 2020-04-16 (Actual); Status verified 2020-04

CONDITIONS: Multicentric Castleman Disease
Keywords: Multicentric Castleman's Disease; Thalidomide, cyclophosphamide and prednisone (TCP regimen); Efficacy; Safety
MeSH Terms: conditions — Multi-centric Castleman's Disease | interventions — Thalidomide; Cyclophosphamide; Prednisone

STUDY DESIGN:
Intervention Model Description: This will be a single center, single arm, phase-II pilot study.
Masking Description: open-labeled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TCP regimen (Experimental): Thalidomide, cyclophosphamide and prednisone （TCP regimen）would be used for newly-diagnosed symptomatic MCD patients
  Interventions: Drug: Thalidomide, cyclophosphamide and prednisone

INTERVENTIONS:
Drug: Thalidomide, cyclophosphamide and prednisone — * Thalidomide: 100mg QN for 1 year; And maintained with 100mg QN for the second year;
  * Cyclophosphamide: 300mg/m2 on Day 1, 8, 15, 22 every month for 1 year;
  * Prednisone: 1mg/kg on Day 1-2, 8-9, 15-16, 22-23 every month for 1 year.
  Other Names: TCP regimen

SUMMARY:
To explore the effectiveness and safety of thalidomide, cyclophosphamide and prednisone (TCP regimen) in newly diagnosed Multicentric Castleman's disease (MCD) patients.

DETAILED DESCRIPTION:
This is a single center, open-labeled , single arm, phase-II pilot study which aims to evaluate the efficacy and safety of thalidomide, cyclophosphamide and prednisone (TCP regimen) in newly diagnosed Multicentric Castleman's disease (MCD) patients.There would be two phases of the study. The treatment and the response evaluation phase will last from the time of enrollment up to 24 months (evaluation will be carried out every 3 months). The follow-up phase to assess for progression of disease will last from 24 months (2 years) to 4 years after enrollment (evaluation will be carried out every 12 months).The total study duration will be 4 years after the last patient starts study medication.

ELIGIBILITY:
* Inclusion Criteria:

  * ≥18 years, all race/ethnic groups in China；
  * Newly diagnosed and previously untreated (patients are allowed to have received oral prednisone for up to 1 week before enrollment) symptomatic MCD patients (symptomatic disease is defined by the presence of clinical symptoms with the NCI-CTCAE grading ≥1 that are attributable to the disease, and for which treatment is indicated);
  * Eastern Cooperative Oncology Group (ECOG) Performance Status ≤2;
  * Clinical laboratory values meeting these criteria at screening: absolute neutrophil count ≥ 1•0 x 109/L, Platelets ≥ 50 x 109/L, Alanine aminotransferase (ALT) within 2•5 x upper limit of normal (ULN); total bilirubin within 2•5 x ULN; estimated glomerular filtration rate (according to MDRD formula) <15ml/min;
  * Women of childbearing potential must agree to use birth control measures during the study and for at least 3 months after receiving the last dose of study agent, and must have a negative pregnancy test at screening period. Men must agree to use birth control measures during the study and for at least 3 months after receiving the last dose of study agent;
  * Informed consent must be signed.
* Exclusion Criteria:

  * age under 18 years;
  * ECOG (eastern cooperative oncology group) status above 2;
  * Immunosuppressive or anti-neoplastic drugs within the last 3 months;
  * serious diseases including malignancy;
  * Plan to have babies within 1 year after enrollment (for women and men), or pregnancy / breast-feeding (for women);
  * Known hypersensitivity to study agents;
  * Active infection requiring systemic treatment;
  * Other severe concurrent disease (eg. uncontrolled diabetes, symptomatic coronary heart disease) that is likely to interfere with study procedures or results, or that in the opinion of the investigator would constitute a hazard for participating in this study;
  * Unwilling or unable to provide informed consent;
  * Unwilling to return for follow-up at PUMCH.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2021-01-01 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang L, Zhao AL, Duan MH, Li ZY, Cao XX, Feng J, Zhou DB, Zhong DR, Fajgenbaum DC, Li J. Phase 2 study using oral thalidomide-cyclophosphamide-prednisone for idiopathic multicentric Castleman disease. Blood. 2019 Apr 18;133(16):1720-1728. doi: 10.1182/blood-2018-11-884577. Epub 2019 Feb 13. PMID 30760451

RESULTS

PARTICIPANT FLOW:
Groups:
- TCP Treatment Group: The newly-diagnosed symptomatic MCD patients received thalidomide, cyclophosphamide and prednisone (TCP ) treatment. The accurate dose of TCP regimen is listed as follows.
  * Thalidomide: 100mg QN for 1 year; And maintained with 100mg QN for the second year;
  * Cyclophosphamide: 300mg/m2 on Day 1, 8, 15, 22 every month for 1 year;
  * Prednisone: 1mg/kg on Day 1-2, 8-9, 15-16, 22-23 every month for 1 year.
Period: Overall Study
Arm/Group | TCP Treatment Group
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | TCP Treatment Group
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 40 [20 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  East Asian | 25
Region of Enrollment [Number; unit: participants]
  China | 25

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Durable Tumor and Symptomatic Response
Description: Durable tumor and symptomatic response is complete response (CR) + partial response (PR). CR: complete disappearance of all measurable and evaluable disease (eg, pleural effusion) and resolution of baseline symptoms attributed to multicentric Castleman's disease, sustained for at least 18 weeks. PR: >=50 percent decrease in sum of the product of the diameters of indicator lesion(s), with at least stable disease in all other evaluable disease in the absence of treatment failure sustained for at least 6 months.
Time Frame: From baseline to the time point when a patient achieves treatment response for 24 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | TCP Treatment Group
Number analyzed (Participants) | 25
Participants | 12

2. Secondary Outcome: Progression-free Survival
Description: Progression-free survival (PFS) is defined as the time to death or treatment failure. Treatment failure is defined as: sustained increase in grade ≥2 disease-related symptoms persisting ≥12 weeks; new disease-related grade ≥3 symptoms; sustained >1 point increase in ECOG-PS persisting for ≥12 weeks; radiological progression; or initiation of another treatment for MCD.
Time Frame: From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | TCP Treatment Group
Number analyzed (Participants) | 25
months | 23.32 [17.22 to 29.42]

3. Secondary Outcome: Overall Survival
Description: Overall survival, defined as the time to patients' death, is measured.
Time Frame: From date of randomization until the date of death from any cause, assessed up to 36 months.
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | TCP Treatment Group
Number analyzed (Participants) | 25
months | 32.16 [28.08 to 36.24]

4. Secondary Outcome: Change in SF-36 Score
Description: SF-36 score is a self-administered scoring system which reflects a patient's general health status. SF-36 contains 8 dimensions, including physical functioning, role physical, role emotional, vitality, mental health, social functioning, bodily pain, and general health. Each dimension ranges from 0 to 100. Higher scores mean better outcome. SF-36 score at baseline was compared with SF-36 score at 24 weeks.
Time Frame: From baseline to 24 weeks after treatment.
Population: Each patient is assessed by SF-36 scoring system, which contains 8 dimensions, including physical functioning, role physical, role emotional, vitality, mental health, social functioning, bodily pain, and general health.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TCP Treatment Group
Number analyzed (Participants) | 25
score on a scale
  physical functioning | 15.1 (6.78)
  role physical | 26.7 (10.53)
  role emotional | 19.6 (10.18)
  vitality | 11.1 (5.75)
  mental health | 8.5 (5.50)
  social functioning | 13.6 (6.70)
  bodily pain | 15.8 (6.19)
  general health | 9.1 (4.78)

5. Secondary Outcome: Number of Participants With Treatment-related Adverse Events as Assessed by CTCAE v4.0 ( ≥1 Grade)
Description: Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 (patients with grades ≥1 would be included)
Time Frame: From initiation of TCP regimen to 3 months after the end of treatment or to time point of the initiation of second line therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | TCP Treatment Group
Number analyzed (Participants) | 25
Participants | 10

6. Secondary Outcome: Number of Participants With Treatment-related Serious Adverse Events as Assessed by CTCAE v4.0 ( ≥3 Grade)
Description: Number of participants with treatment-related serious adverse events as assessed by CTCAE v4.0 (patients with grades ≥3 would be included)
Time Frame: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | TCP Treatment Group
Number analyzed (Participants) | 25
Participants | 2

ADVERSE EVENTS:
Time Frame: Safety data were collected until 30 days after the last dose of study drugs, except for secondary primary malignancies (which were assessed throughout the duration of follow-up, up to 4 years). Secondary primary malignancies were assessed throughout the duration of follow-up, up to 3 years.
Arm/Group | TCP Treatment Group
All-Cause Mortality (participants affected / at risk) | 3/25
Serious Adverse Events (participants affected / at risk) | 2/25
Other Adverse Events (participants affected / at risk) | 10/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TCP Treatment Group (N=25)
Pulmonary infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Skin rash (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TCP Treatment Group (N=25)
constipation (Gastrointestinal disorders) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-01): https://cdn.clinicaltrials.gov/large-docs/05/NCT03043105/Prot_SAP_000.pdf